CLINICAL TRIAL: NCT00602823
Title: Ex Vivo Monocyte and Lymphocyte Stimulation Tests and Genomic Study for the Prediction of Efficacy and Adverse Effects of CD11a Monoclonal Antibodies(Raptiva)
Brief Title: Genomic Study for the Prediction of Efficacy and Adverse Effects of CD11a Monoclonal Antibodies(Raptiva)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561701002; 9561701002
Record Dates: First submitted 2007-03-22; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2006-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

SUMMARY:
The pathogenesis of psoriasis has evolved from epidermal hyperproliferation to immune dysregulation in recent years. A Th1 cytokine profile is universally found is psoriasis. Biologics targeting the immune system have become the focus of study. Raptiva (Efalizumab) is one of biologics indicated for the treatment of psoriasis, and is the first biologic approved for use in psoriasis in the EU (EMEA). In USA, it is the second biologic drug (after Amevive) for psoriasis. Raptiva is a humanized chimeric antibody of CD11a (LFA-1), which blocks the interaction of CD11and ICAM-1, thus preventing lymphocyte trafficking. It is used for moderate to severe chronic plaque type psoraisis. The first clinical trial of Raptiva in Asians iscurrently done in the department of Dermatology, National Taiwan University Hospital and the incidence of psoriatic arthritis (either de novo or aggravation of preexisting psoriatic arthritis) is significantly higher than previously reported in Western countries（30％ versus 7%，and personal communication with doctors in Hong-Kong and Singapore also reveals a similar safety profile. It seems likely that a racial difference is present. Monocytes play a central role in the pathogenesis of psoriatic arthritis. It is thus intriguing to study the pathogenesis of Raptiva-induced aggravation of psoriatic arthritis by comparing the difference of monocyes response in the presence of Raptiva between patients with and without Raptiva-induced psoriatic arthritis. In further study, the CD11a genomic polymorphism will also be investigated. The suudy can provide us with important information on how a novel monoclonal antibody like Raptiva can have both therapeutic and detrimental actions on psoriasis. The short term benefit of the study will be in pharmacogenomics and pharmacoeconomics, finding the best candidates for the expensive drug. The long term goal will be the clarification of the pathogenesis of psoriasis and psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-02; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: TSEN-FANG Tsai, MD, Study Chair — TSEN-FANG Tsai